CLINICAL TRIAL: NCT02917304
Title: A Multicenter, Open-label, Single Arm Study to Evaluate the Immunological Efficacy and Safety of GC3110A. Administered Intramuscularly in Healthy Subjects Aged 65 Years and Older
Brief Title: A Study to Evaluate the Efficacy and Safety of GC3110A in Healthy Subjects Aged 65 Years and Older
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GC3110A_ED_P3
Record Dates: First submitted 2016-09-26; First posted 2016-09-28 (Estimated); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Influenza, Human
Keywords: Quadrivalent Influenza Vaccines
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- GC3110A vaccine group (Experimental): Participants administered a single dose of GC3110A(Quadrivalent Influenza Vaccine).
  Interventions: Biological: GC3110A vaccine

INTERVENTIONS:
Biological: GC3110A vaccine — 0.5mL, Intramuscular
  Other Names: GC3110A

SUMMARY:
The purpose of this study is to evaluate immunological efficacy and safety of GC3110A among healthy adults over 65 years of age.

DETAILED DESCRIPTION:
Adults over 65 years of age will be once administered GC3110A(Quadrivalent influenza vaccine).

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults aged 65 years and older
* Informed consent form has been signed and dated
* Able to comply with the requirements of the study

Exclusion Criteria:

* Known systemic hypersensitivity to eggs, chicken proteins, or any of the vaccine components
* Personal history of Guillain-Barre syndrome(GBS)
* Subjects with severe chronic disease who are considered by investigator to be ineligible for the study
* Subjects who received a vaccination within 28 days before enrollment or who are scheduled for another vaccination during the study
* Immunocompromised subjects with immunodeficiency disease or subjects receiving immunosuppressive or immunomodulating therapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 274 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2016-12-02 (Actual); Study Completion 2017-05-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants Achieving Pre-defined Seroconversion Before and following vaccination | Day 0 (Pre-Vaccination) and Day 21 (Post-Vaccination)
  Percentage of Participants Achieving Pre-defined Seroconversion Before and following vaccination
Percentage of Participants Achieving Pre-defined Seroprotection Before and following vaccination | Day 0 (Pre-Vaccination) and Day 21 (Post-Vaccination)
  Percentage of Participants Achieving Pre-defined Seroprotection Before and following vaccination

SECONDARY OUTCOMES:
Geometric Mean Titer and Geometric Mean Titer Ratios of Antibodies to the GC3110A Before and Following Vaccination | Day 0 (Pre-Vaccination) and Day 21 (Post-Vaccination)
  Geometric Mean Titer and Geometric Mean Titer Ratios of Antibodies to the GC3110A Before and Following Vaccination

CONTACTS AND LOCATIONS:
Locations (10):
- South Korea (10):
  - The Catholic Univ. of Korea Daejeon St.Mary's Hospital, Daejeon
  - Soon Chun Hyang University Bucheon Hospital, Gyeonggi-do
  - The Catholic Univ.of Korea Bucheon St.Mary's Hospital, Gyeonggi-do
  - The Catholic Univ.of Korea Uijeongbu St.Mary's Hospital, Gyeonggi-do
  - EWHA woman's university mokdong hospital, Seoul
  - KyungHee University Medical Center, Seoul
  - Soon Chun Hyang University Seoul Hospital, Seoul
  - The Catholic Univ. of Korea Incheon St.Mary's Hospital, Seoul
  - The Catholic Univ.of Korea Seoul St.Mary's Hospital, Seoul
  - The Catholic Univ.of Korea Yeouido St.Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No